CLINICAL TRIAL: NCT01767402
Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the Pneumococcal Protein PhtD Vaccine Without or With Adjuvant, Administered at 2 Different Concentrations According to a 0-2 Month Schedule, in Healthy Adults
Brief Title: Study to Evaluate Safety, Reactogenicity and Immunogenicity of the Pneumococcal Protein PhtD Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 100417
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Pneumococcal Disease
Keywords: Safety; Pneumococcal Infections; Immunogenicity; PhtD vaccine; Healthy adults; Reactogenicity
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- PhtD Group 1 (Experimental): Subjects will receive PhtD vaccine formulation 1 without any adjuvant.
  Interventions: Biological: PhtD vaccine with/without adjuvant
- PhtD Group 2 (Experimental): Subjects will receive adjuvanted PhtD vaccine formulation 2.
  Interventions: Biological: PhtD vaccine with/without adjuvant
- PhtD Group 3 (Experimental): Subjects will receive adjuvanted PhtD vaccine formulation 3.
  Interventions: Biological: PhtD vaccine with/without adjuvant
- PhtD Group 4 (Experimental): Subjects will receive adjuvanted PhtD vaccine formulation 4.
  Interventions: Biological: PhtD vaccine with/without adjuvant
- PhtD Group 5 (Experimental): Subjects will receive adjuvanted PhtD vaccine formulation 5.
  Interventions: Biological: PhtD vaccine with/without adjuvant
- 23 PPV Group (Active Comparator): Subjects will receive the Pneumovax 23TM vaccine and NaCl.
  Interventions: Biological: Pneumovax 23TM; Biological: NaCl

INTERVENTIONS:
Biological: PhtD vaccine with/without adjuvant — Two doses of different formulations of PhtD vaccine administered intramuscularly in the deltoid region of the right arm at month 0 and month 2.
  Arms: PhtD Group 1; PhtD Group 2; PhtD Group 3; PhtD Group 4; PhtD Group 5
Biological: Pneumovax 23TM — One dose of Pneumovax 23TM vaccine administered intramuscularly in the deltoid region of the right arm at month 0.
  Arms: 23 PPV Group
Biological: NaCl — One dose administered intramuscularly in the deltoid region of the right arm at month 2.
  Arms: 23 PPV Group

SUMMARY:
The purpose of this study is to examine the safety, reactogenicity and immunogenicity of the GlaxoSmithKline (GSK) Biologicals candidate pneumococcal vaccine containing PhtD in healthy elderly population aged 18-45 years of age.

DETAILED DESCRIPTION:
The safety profile of the PhtD vaccine will be assessed in comparison to a comparator vaccine (Pneumovax 23TM). In order to further increase the immune response to vaccination, a novel adjuvant system will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 18 and 45 years at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential, i.e., either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period or participation to another pharmaceutical/vaccine study.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Use of any anticoagulants.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 2 weeks of the first dose of vaccines.
* Previous vaccination against Streptococcus pneumoniae.
* Bacterial pneumonia within 3 years prior to 1st vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Current serious neurologic or mental disorders.
* Inflammatory processes such as known chronic active infections.
* All malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders diagnosed or treated actively during the past 5 years.
* History of administration of an experimental vaccine containing 3-deacylated Monophosphoryl Lipid A (MPL) or Quillaja saponaria 21 (QS21).
* Acute disease at the time of enrolment. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., Oral temperature <37.5°C or Axillary temperature <37.5°C.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, at the discretion of the investigator.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or intravenous drug abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2003-10; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship of any solicited local and general signs and symptoms | During a 7-day follow up period (i.e. Days 0-6) after each vaccine dose
Occurrence, intensity and relationship to vaccination of unsolicited local and general signs and symptoms | During a 30-day follow up period (i.e. Days 0-29) after each vaccine dose
Occurrence of all serious adverse events (SAEs) | During the 12 months of the study
Anti-PhtD antibody concentration in all vaccine groups (measured by ELISA) | One month after the first injection
Anti-PhtD antibody concentration in all vaccine groups (measured by ELISA) | One month after two injections

SECONDARY OUTCOMES:
Number and percentage of subjects with normal or abnormal values, for biochemical assessments and for hematological analysis | At month 0, 1, 3 and 12
Anti-PhtD antibody concentration in all groups (measured by ELISA) | At 12 months after the first vaccination
Anti-PhtD antibody avidity (measured by ELISA) | At month 0, 1, 3 and 12
Evaluation of protection afforded by passive transfer of anti PhtD antibodies sera pooled from all individuals (passive transfer mice model assay) | At month 0, 1, 3 and 12
Frequency of PhtD-specific plasma cells generated by in vitro cultivated memory B-cells in a subset of subjects (measured by B-cell ELISPOT) | At month 0, 3 and 12
Frequency of CD4 and/or CD8 T cells that produce cytokines IL-2, IL-4, IFNg, CD40L and/or GM-CSF, upon PhtD re-stimulation in vitro, to evaluate the T-cell response, in a subset of subjects (measured by intracellular cytokine cytometry) | At month 0, 3 and 12
Anti-polysaccharide total gamma class immunoglobulin (IgG) concentration in the 23 valent Polysaccharide Pneumococcal Vaccine(23 PPV) group for 11 serotypes (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, 23F) (ELISA) | At month 0, 1 and 12
Opsonophagocytic activity titers in the 23 PPV group for 11 serotypes (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, 23F (OPA assay) | At month 0, 1 and 12
Frequency of polysaccharide(PS)-specific plasma cells generated by in vitro cultivated memory B-cells in the 23 PPV group in a subset of subjects (measured by B-cell ELISPOT) | At month 0, 1 and 12
Circulating serum cytokines Interferon-gamma (INFγ) and Tumor necrosis factor-alpha (TNFα) content in all groups (measured by ELISA) | At Day 0, 1, 60 and 61

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Leroux-Roels I, Devaster JM, Leroux-Roels G, Verlant V, Henckaerts I, Moris P, Hermand P, Van Belle P, Poolman JT, Vandepapeliere P, Horsmans Y. Adjuvant system AS02V enhances humoral and cellular immune responses to pneumococcal protein PhtD vaccine in healthy young and older adults: randomised, controlled trials. Vaccine. 2015 Jan 15;33(4):577-84. doi: 10.1016/j.vaccine.2013.10.052. Epub 2013 Oct 29. PMID 24176494